CLINICAL TRIAL: NCT06867458
Title: Steriwave ICU Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: Ondine Biomedical Inc. (Industry); Royal Columbian Hospital Foundation (Other)
Responsible Party: Principal Investigator, Steve Reynolds, Critical Care Physician, Fraser Health
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2024142
Record Dates: First submitted 2025-03-01; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Ventilator Acquired Pneumonia; Hospital Acquired Pneumonia; Hospital Acquired Infections; Nasal Decolonization of Staphylococcus Aureus
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia

STUDY DESIGN:
Intervention Model Description: The pilot study will take place over four months at the Royal Columbian Hospital (RCH) Intensive Care Units. All patients who meet inclusion/exclusion criteria will be enrolled via a waived consent procedure. The first two months will constitute the control period before the aPDT intervention is introduced into the unit. All patients enrolled in the study will receive a nasal swab upon ICU admission, and once every four days during their stay. Following the control period, the intervention period will commence with the introduction of the aPDT device to all eligible patients. Nasal decolonization procedures will be administered every other day. Patients will undergo one follow-up visit at 4 days post ICU discharge.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): The first two months will constitute the control period before the aPDT intervention is introduced into the unit. No nasal decolonization procedures (current standard of care) will take place at this time. All patients enrolled in the study will receive a nasal swab upon ICU admission, and once every four days during their stay.
- Intervention Arm (Experimental): Nasal decolonization procedures will be administered every other day. Just as during the intervention period, a nasal swab will be administered every four days to assess the microbiology of the nose prior to the scheduled nasal decontamination treatment
  Interventions: Device: Antimicrobial photodynamic therapy (aPDT) nasal decolonization device

INTERVENTIONS:
Device: Antimicrobial photodynamic therapy (aPDT) nasal decolonization device — aPDT is a technique that employs a specific wavelength of light to activate a photosensitizer substance. Once activated, this photosensitizer reacts with surrounding molecules to produce radicals and reactive oxygen species. When activated in the presence of microorganisms, these molecules serve to disrupt membrane structure and protein cross-linking, leading to their death.
  Arms: Intervention Arm

SUMMARY:
This is a single-center, non-blinded, prospective, pilot study enrolling patients admitted to the critical care unit at Royal Columbian Hospital. This study investigates the effects of universal nasal decolonization using antimicrobial photodynamic therapy (aPDT) on the prevention of hospital-acquired pneumonia (HAP), ventilator-acquired pneumonia (VAP), and hospital-acquired bloodstream infection (BSI) in this patient population.

Main Objectives include:

* To determine whether a large, multi-center RCT of this protocol is feasible
* To determine baseline rates of VAP, HAP, and ICU-acquired BSI
* To gather preliminary efficacy data regarding VAP, HAP, and ICU-acquired BSI prevention using universal aPDT nasal decolonization
* To gather preliminary microbiological data on the effect of universal aPDT procedures on nasal carriage of various microoganisms in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients 19 years and above
* Expected length of ICU stay >48 hrs

Exclusion Criteria:

* Pregnant/breastfeeding individuals
* Allergy to methylene blue and/or chlorhexidine gluconate, or unknown allergy status
* Nasal or facial trauma that limits access to the nose
* Inability for the patients to tolerate or comply with treatment, as determined by their treating physician
* Patient, TSDM or MRP declines participation
* Co-enrolment with other research studies will be considered in an individual basis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
Protocol Adherance | Entire study duration- 4 months
  During each day of the study, members of the research team will track adherence to the nasal swab and nasal decolonization procedures (during the intervention phase) for all patients enrolled in the study. A standardized checklist will be developed and used to track protocol adherence.

SECONDARY OUTCOMES:
Change in nasal bacterial load | Entire study duration- up to 4 months
  Change in nasal bacterial load will be measured by a decrease in semi-quantitative (1+ to 4+) growth on blood agar plates. Nasal swab samples will be collected on every 4th day of the patients ICU stay, with one additional swab collected 4-days post- ICU discharge, should the patient remain hospitalized at the same institution.
Preliminary Microbiology Data | Entire study duration- up to 4 months
  Change in CPO, MRSA, MSSA, and MDR gram-negative (Pseudomonas and SPACE organisms) carriage rates. Nasal swab samples will be collected on every 4th day of the patients ICU stay, with one additional swab collected 4-days post- ICU discharge, should the patient remain hospitalized at the same institution.
HAP incidence | Entire study duration- up to 4 months
  HAP will be diagnosed according to the Fraser Health Antimicrobial Stewardship Program (ASP) Hospital Acquired Pneumonia definition. This document defines a HAP event as "pneumonia that occurs 48 hours or more after admission and was not present at the time of admission." Whether or not a patient is diagnosed with pneumonia will be adjudicated according to the January 2024 National Health and Safety Network (NHSN) diagnosis algorithm. Additionally, if the patients treating physician diagnoses the patient with HAP, this will be considered sufficient to include as a study outcome. Data needed to adjudicate this outcome will be collected from patient charts by members of the research team. This data will be compiled for analysis by the same committee as noted above.
VAP incidence | Entire study duration- up to 4 months
  As above, VAP will also be diagnosed according to Fraser Health ASP Ventilator- Associated Pneumonia definition, as a "pneumonia that occurs 48 hours after endotracheal intubation." The causative organism must be different than an organism present form any index infection prior to the ICU stay. The presence of pneumonia will be similarly adjudicated according to the NHSN diagnosis algorithm. Any mention of VAP in the physicians progress notes will also be deemed sufficient for study outcomes.
ICU-acquired BSI incidence | Entire study duration- up to 4 months
  ICU-acquired BSI will be diagnosed in accordance with the CDC National Healthcare Safety Network BSI definition from January 2024, described as "a laboratory confirmed bloodstream infection that is not secondary to an infection at another site". In order for the infection to be considered ICU-acquired, the patient must have tested for a new pathogen (that is not a common commensal) 48 hours after their ICU admission date. We will consider a BSI from any cause as contributing to this outcome.
Ability to adjudicate HAP occurrence effectively | Entire study duration- 4 months
  We will consider adjudication effective if we are able to complete the process using data collected in the study CRFs within 30 days of protocol completion.
Ability to adjudicate VAP occurrence effectively | Entire study duration- 4 months
  We will consider adjudication effective if we are able to complete the process using data collected in the study CRFs within 30 days of protocol completion.
ICU Readmission | Entire study duration- 4 months
  Number of patients re-admitted to the ICU during the 4-day follow-up
LOS- Hospital | Entire study duration- 4 months
  Hospital length of stay (days)
LOS- ICU | Entire study duration- 4 months
  ICU length of stay (days)
In-hospital mortality up to 60 days post intervention | One time measurement, 60 days post- ICU admission
  At 60 days post-ICU admission, we will record information about patient death as it is available from the same visit on the EMR. We will not gather data on any information that occurred outside of the immediate study visit. We will not contact participants who have been discharged from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, Principal Investigator — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data set may be available upon reasonable request.